CLINICAL TRIAL: NCT03667313
Title: Prospective Randomised Study Comparing Efficacy of Treatment Coronary In-stent Restenosis Using Sirolimus-Eluting and Iopromide-Coated Paclitaxel-Eluting Balloon Catheters
Brief Title: Treatment of In-Stent Restenosis 2 Study
Acronym: TIS2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FNO-TIS 2
Record Dates: First submitted 2018-09-10; First posted 2018-09-12 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-12

CONDITIONS: Coronary Restenosis
Keywords: in-stent restenosis; sirolimus-; paclitaxel-eluting balloon
MeSH Terms: conditions — Coronary Restenosis | interventions — BEP protocol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sirolimus-eluting balloon (SEB) (Experimental): treatment of bare-metal (BMS) or drug-eluting in-stent restenosis (DES-ISR) with SEB
  Interventions: Combination Product: sirolimus-eluting balloon (SEB) MagicTouch
- paclitaxel-eluting balloon (PEB) (Active Comparator): treatment of BMS- or DES-ISR with PEB
  Interventions: Combination Product: paclitaxel-eluting balloon (PEB) Sequent Please

INTERVENTIONS:
Combination Product: sirolimus-eluting balloon (SEB) MagicTouch — Patients with coronary in-stent restenosis treated with sirolimus-eluting balloon
  Other Names: MagicTouch
  Arms: sirolimus-eluting balloon (SEB)
Combination Product: paclitaxel-eluting balloon (PEB) Sequent Please — Patients with coronary in-stent restenosis treated with paclitaxel-eluting balloon
  Other Names: Sequent Please
  Arms: paclitaxel-eluting balloon (PEB)

SUMMARY:
The aim of this study is to compare the efficacy of sirolimus-eluting balloon catheters (SEB) and iopromide-coated paclutaxel-eluting balloon catheters (PEB) in the treatment of bare metal (BMS) - or drug-eluting stents restenosis (DES-ISR).

DETAILED DESCRIPTION:
Current therapy for in-stent restenosis (ISR) is based on the drug-eluting stents (DES) or drug-eluting balloon catheters (DEB). In clinical practice, paclitaxel is used as an effective antiproliferative agent loaded into DEB (paclitaxel-eluting balloon catheters; PEB).

In contrast to paclitaxel, sirolimus is difficult to deliver on the balloon surface, due to insufficient tissue uptake and shorter tissue retention of limus drugs. It was found that phospholipid-encapsulated sirolimus nanoparticles could be used for coating balloon catheters to provide efficient drug transfer to vessel wall with high tissue concentration.

This prospective randomized non-inferiority study compares the efficacy of new sirolimus-eluting balloon catheters (SEB) and iopromide-coated paclutaxel-eluting balloon catheters (PEB) in the treatment of bare metal (BMS) - or drug-eluting stents restenosis (DES-ISR).

The primary end-point is in-segment late lumen loss (LLL) at 12 months as measured by quantitative coronary angiography (QCA).

Secondary end-points are the incidence of binary ISR (˃50% DS) and the overall incidence of 12-month major adverse cardiac events (MACE; cardiovascular death, non-fatal acute myocardial infarction [AIM], or target vessel revascularization [TVR]).

ELIGIBILITY:
Inclusion Criteria:

* patients with BMS- or DES-ISR (˃50% diameter stenosis; DS)
* ≥18 years of age
* willing to sign an Informed consent

Exclusion Criteria:

* concomitant diseases with an expected survival time of less than 12 months
* or that limited the possibility of control coronary aniography (e.g., advanced renal failure).
* impossibility of long-term (6 months) dual antiplatelet treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Late lumem loss (LLL) | 12-month
  the diference between post-intervention mimimal lumen diameter (MLD) and 12-month MLD

SECONDARY OUTCOMES:
repeated binary restenosis | 12-month
  recurrence of stenosis ≥50%
major adverse cardiac events (MACE) | 12-month
  cardiovascular death, non-fatal acute myocardial infarction [AIM], or target vessel revascularization [TVR]

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiovascular Department of University Hospital, Ostrava, Czechia

REFERENCES:
- [Derived] Pleva L, Kukla P, Kovarnik T, Zapletalova J. Comparing the Efficacy of Sirolimus and Paclitaxel-Eluting Balloon Catheters in the Treatment of Coronary In-Stent Restenosis: A Prospective Randomized Study (TIS 2 Study). Circ Cardiovasc Interv. 2025 May;18(5):e014677. doi: 10.1161/CIRCINTERVENTIONS.124.014677. Epub 2025 Apr 2. PMID 40171676